CLINICAL TRIAL: NCT00715052
Title: The Effect of Hyperbaric Oxygen Therapy on Patients Suffering From Neurologic Deficiency Due Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Shai Efrati, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HBOtbi1
Record Dates: First submitted 2008-07-14; First posted 2008-07-15 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2008-10

CONDITIONS: Neurologic Deficiency; Traumatic Brain Injury
Keywords: neurologic deficiency due traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 40 consecutive one hour treatments at 1.5 ATA with 100% O2
  Interventions: Procedure: Hyperbaric Oxygen Therapy (HBOT)
- 2 (No Intervention)

INTERVENTIONS:
Procedure: Hyperbaric Oxygen Therapy (HBOT) — 40 consecutive one hour treatments at 1.5 ATA with 100% O2
  Arms: 1

SUMMARY:
Traumatic brain injuries (TBI) are a major cause of morbidity and mortality worldwide. Due to improvements in emergency medical care, transportation and specialized trauma facilities, the number of people surviving TBI with impairment has significantly increased in recent years. The long term cognitive sequelae, which are often not visible persist far beyond the resolution of the obvious physical disabilities. This combined with the relatively low awareness of the general public has designated TBI as the "silent epidemic" (TBI CDC 2006). Hyperbaric oxygen therapy (HBOT) has been suggested as a possible treatment modality for these cases and preliminary studies are promising.

The purpose of this study is to evaluate the effectiveness of HBOT in the treatment of chronic mild traumatic brain injuries (mTBI). Sequential SPECT scans of the brain and neurocognitive testing will be used to evaluate cerebral blood flow (CBF) response, cognitive and functional improvement following treatment.

DETAILED DESCRIPTION:
INTRODUCTION Traumatic brain injuries (TBI) are a major cause of morbidity and mortality worldwide. Due to improvements in emergency medical care, transportation and specialized trauma facilities, the number of people surviving TBI with impairment has significantly increased in recent years. The long term cognitive sequelae, which are often not visible persist far beyond the resolution of the obvious physical disabilities. This combined with the relatively low awareness of the general public has designated TBI as the "silent epidemic" (TBI CDC 2006). Hyperbaric oxygen therapy (HBOT) has been suggested as a possible treatment modality for these cases and preliminary studies are promising.

The purpose of this study is to evaluate the effectiveness of HBOT in the treatment of chronic mild traumatic brain injuries (mTBI). Sequential SPECT scans of the brain and neurocognitive testing will be used to evaluate cerebral blood flow (CBF) response, cognitive and functional improvement following treatment.

Traumatic brain injuries (TBI) Traumatic brain injuries are a major cause of morbidity and mortality leading to major long term consequences on both a personal and national level with an estimated 5.3 million Americans suffering from permanent TBI related disabilities (24).The prevalence of traumatic brain injury in the United States is estimated to be approximately 1.5 million individuals per year (24,25). This however does not include those individuals who did not receive care in a facility included in national surveillance systems or received no medical care at all and thus probably significantly underestimates the actual number of TBI victims. The 2006 NIH consensus states a prevalence of 2.5 - 6 million people per year suffer form TBI(23).

Due to improvements in emergency medical care, transportation and specialized trauma facilities, the number of people surviving TBI with impairment has significantly increased in recent years. The long term consequences of TBI are vast, affecting a large number of people with a substantial effect on the patients themselves, their families and society as a whole. These injuries also impart a significant economic burden on those involved, both personally and as a society. Approximately 80,000 - 90,000 individuals suffer from long term disabilities annually, and the estimated costs including both direct medical care and indirect expenses such as lost earning potential were over 60 million dollars in 2001 in the US (28).

The long term sequelae of TBI may include impairment of the individuals physical, cognitive and psychosocial functioning. The neurological consequences are numerous and complex affecting various sites and functions. Sensory, motor and autonomic systems may all be affected and symptoms may include headaches, seizures, visual defects, movement disorders and sleep disorders. The cognitive consequences likewise are broad and varied. Amongst the symptoms most commonly noted are memory deficits and problems with attention and concentration. There may be impaired executive function, problem solving abilities and language difficulties as well as problems with planning, information processing, judgment and insight. While some of these symptoms may be apparent immediately after the injury, others may present days, weeks or months after the initial trauma(Kushner,24). Moreover, there can be vast fluctuations and changes in the severity and presentation over time.

Another realm of difficulties resulting from TBI includes behavioral, emotional and psychological impairments. There can be vast personality changes including loss or decreased ability to initiate responses and activities, disinhibition, impulsivity, aggressive behaviors - both verbal and physical, and changes in sexual behavior. Personality and mood disorders may appear and depression, anxiety and changes in emotional control are often noted after TBI.(23) The social consequences may also be widespread and often devastating. There is an increased incidence of divorce, chronic unemployment, suicide and substance abuse following TBI. Even in the more chronic stages as the patient is in the recovery stage, the increased demands placed on him in the workplace or upon undertaking new tasks may uncover problems with executive functions and planning abilities that had as of yet been unnoticed.

These problems and the burden of caring for these individuals on a long term basis place cumulative strains on the family and their support network. Family members and care givers report an increased occurrence of depression, anger and social isolation. These combine to result in disrupted family functioning and relationships and these problems may persist or worsen with time.(24)

HBO for TBI Hyperbaric Oxygen Therapy (HBOT) has been in use since the 1930's when it was initially used for decompression sickness. Shortly thereafter physicians started usingHBOT for a variety of other conditions. The use of HBOT for neurological indications started in the early 1960s with the work by Smith et al showing its protective effect in cerebral ischemia and that of Saltzman showing effectiveness in stroke patients.(Jain) HBOT is the inhalation of 100% oxygen at pressures exceeding 1 atmospheres absolute (ATA) in order to enhance the amount of oxygen dissolved in the blood and body fluids, thereby allowing for increased oxygen delivery to the tissues. The mechanism by which HBOT is thought to improve the outcome of brain injury is multifaceted.

The Neubauer and Walker(2000) theory postulates that HBOT improves cerebral metabolism by improving functioning of the dormant neurons and stimulating axonal growth (10). Zhang et al suggest that potential targets of oxygen therapy include prevention of apoptosis, inhibition of neuroinflammation and BBB damage (Zhang pathophysiology 2005,Rossignol). There is stimulation of angiogenesis and neovascularization, as well as direct effects on blood vessels in the brain, and maintenance of BBB integrity. (1((5-12)),20) . Similarly, SPECT scans have demonstrated a positive effect on the cerebral blood flow (CBF) in the damaged brain following HBOT (2,8,10,16,19,17,neubauer HBOT of closed head,20,). HBOT also brings about improved neurocognitive functioning in patients suffering from chronic brain injury. (14,9,6,13,20,21).

Under normobaric conditions, the amount of oxygen dissolved in the blood is only 0.3 ml/dl. At 1.5 ATA this amount increases 10 fold to 3.2 ml/dl. Using an animal model of brain injured mice Daughrty et al (rockswall 9) found a 250% increase in the local brain tissue oxygen levels between 100% oxygen administered at 1 ATA (103 mmHg) as opposed to that given at 1.5 ATA (247 mmHg). This seems to suggest that the this dissolved O2 is more readily available to the brain tissue than hemoglobin bound oxygen (20). Additionally, work by several investigators seems to indicate that HBOT allows for more efficient use of baseline oxygen levels by injured brain tissue following treatments, which in turn leads to a positive persistent affect on this tissue (20).

It has been theorized that following brain injury from any cause, there is an area of "idling neurons" in the ischemic penumbra zone which are still viable and potentially salvageable if given the right treatment. This area consists of dormant neurons between the areas of dead tissue and the unaffected healthy tissue surrounding it. .(2,16,17,18,19,jain,22). There appears to be sufficient oxygen available to these cells to maintain cell life and ion pump mechanisms, but not enough to generate action potentials and allow them to act as functioning neurons (17,19).

The hyperoxia from HBOT causes vasoconstriction of the cerebral blood vessels which has been shown to cause a decrease in brain edema and ICP (11,13,6,7,12 fr rockswald ). This vasoconstriction does not appear to have any harmful affect on the brain tissue due to the greatly increased oxygen availability to the tissue. There is also a beneficial effect effect on the BBB, evidence by reduce post ischemic BBB permeability defect (jaine,veltkamp, rockswald 52,55,63).

There are well documented animal models of TBI and a growing body of literature using HBOT on these animal models verifying the above stated hypotheses and findings.

Sun et al demonstrated improved penumbral oxygenation following HBO treatment in focal ischemia using an animal model by measuring both extrinsic and intrinsic markers of hypoxia (SUN). Harch et al used a rat model of TBI to evaluate HBO effects on spatial learning and memory, as well as it's affect on blood vessel density. After receiving a unilateral cortical contusion, Long-Evans rats were tested in the Morris Water Task (MWT) 31-33 days post injury. The rats were divided into an untreated control group, a sham-treated normobaric air group and an HBO group which received 80 bid treatments of HBO at 1.5 ATA/90 mins. The rats were subsequently retested in the MWT and then euthanized. Blood vessel density was measured bilaterally in the hippocampus and correlated with the MWT performance. The HBOT caused a significant increase in the hippocampal vascular density (p< 0.001) and an associated significant improvement in spatial learning (p< 0.001) compared to the control groups. Similarly, the increased vascular density and the improved MWT in the HBOT group were highly correlated (p<0.001). (11)

SPECT for investigation and follow up Single photon emission CT (SPECT) scans have been found to be effective in evaluating post traumatic lesions in mTBI patients and are useful as a means of follow up of recovery.

In a prospective study to evaluate the usefulness of SPECT scans in the diagnosis of patients with mTBI and it's correlation with common clinical symptoms such as post concussion syndrome (PCS), post traumatic amnesia (PTA) and loss of consciousness (LOC), Gawda et al found perfusion abnormalities in 63% of the patients. This as opposed to positive CT findings in only 34% of these patients. In adults, the frontal lobe was most commonly affected whereas the temporal lobes were more likely to be involved in children. The SPECT scan was found to be more sensitive than CT in patients presenting with LOC, PTA and PCS (14).

Jacobs et al evaluated the predictive value of SPECT scans for clinical outcome of 136 mTBI patients in a prospective study. None of the patients had abnormal findings on CT. All patients underwent initial SPECT scans and CT scans within 4 wks of the trauma. Follow up evaluations were performed 3, 6, and 12 months post injury. All patients with abnormal SPECT studies or deteriorating clinical findings had follow up SPECT scans performed at the subsequent time of evaluation.

The initial SPECT was positive in 54% of the patients with a gradual decrease in the number of positive scans over time. The clinical normalization occurred more rapidly than did the normalization of the imaging studies. The SPECT was shown to have high sensitivity and negative predictive value from 3 months post injury onward so that a negative early SPECT is a reliable criteria in the exclusion of clinical sequelae. A positive initial SPECT scan did not exclude a positive clinical outcome, however, a positive SPECT scan at 12 months post injury was a reliable predictor for clinical outcome (13). Golden et al showed improved blood flow as measured by sequential SPECT studies in 50 patients with chronic neurological disorders (10).

SHI Xiao -yan presented a large study of 310 patients in which the effect of HBOT on CBF as well as the usefulness of SPECT in the diagnosis and assessment of neurocognitive disorders following TBI was examined. Pre and post treatment scans were compared and the percent of positive initial SPECT scans was substantially higher than those found with CT alone (81.3% vs. 15.2%). Following HBOT 63.5% of the SPECT scans had normalized concomitant with marked improvement of the clinical symptoms of headache, dizziness, poor concentration and poor memory. An additional 36.5% of the initial positive SPECT scans showed between 33-66% improvement in CBF along with clinical improvement as well.

Proposed Study Design Sixty consenting TBI patients at any age who are at least one year post injury with stable cognitive deficits will be recruited. Any patient with previous neurological deficits, head trauma or substance abuse will be excluded as well as anyone with any contraindications for HBOT. All patients or their trustees will sign written informed consent before their inclusion and the study protocol will be approved by the local Helsinki committee.

Patients will be excluded if they will have one of the following criteria:

1. Had been treated with HBOT for any indiction prior to their inclusion.
2. Have any other indication for HBOT
3. Chest pathology incompatible with pressure changes
4. Inner ear disease
5. Patients suffering from claustrophobia.
6. Inability to give written informed consent by the patient or his trustee. A complete history including medical and concurrent medications will be recorded. Patients will undergo evaluation of activities of daily living (ADL), physical examination, neurocognitive testing and SPECT scan will be performed at baseline. Mild traumatic brain injury will be defined according to the 1993 American Congress of Rehabilitation Medicine definition as a head trauma with loss of consciousness lasting less than 30 minutes, a Glasgow Coma Score (GCS) score of 13 or more, and posttraumatic amnesia lasting less than 24 hours. (Kay et al).

The patients will be randomly assigned to two groups. Group I will initially receive 40 consecutive HBOT treatments and Group II no HBOT treatment. At the end of this first phase of approximately two months, both groups will be revaluated with a second SPECT scan and neurocognitive testing. There will then be a cross over of the two groups and Group II (previously none treated) will receive HBOT treatment while Group I (previously treated) will not receive any further treatments. Again at the end of this second phase there will be follow up SPECT scans and neurocognitive testing for both groups. Additionally at the end of each phase there will be a detailed questioner assessing adverse effects and evaluating any changes in ADL.

There will be an evaluation of the results after the first phase comparing the differences between the treated and non treated groups as well as allowing for evaluation of any spontaneous changes occurring in the non treated group due to the passage of time or a learning curve for the cognitive evaluation.

Following completion of the second phase there will be another evaluation of the results comparing the effect of HBOT on Group II as compared to their baseline as well as evaluating whether the effects seen in Group I are maintained after two months with no treatment.

The HBOT treatment will consist of 40 consecutive one hour treatments at 1.5 ATA with 100% O2 in either a multiplace or monoplace unit per patient preference. The treatments will be given once daily five times a week.

Cognitive evaluation

Statistical analysis This is a pilot randomized crossover study. The sample size of 30 patients in each subgroup (total 60 patients) in the post ischemic stroke as well as in the post hemorrhagic stroke was determined in order to achieve 90% power based on the following assumption related to the expected change in neurologic evaluation: mean difference between the groups of at least 25% with drop rate of 16% and alpha 5% before the cross match period.

Statistical analysis will be performed using the statistical software SPSS-version 13. Parametric data will be expressed as means ± standard deviations and compared by one way ANOVA. Non-parametric data will be compared using Kolmogorov-Smirnov test. Differences between the results yielding p values less than 0.05 (p<0.05) will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* TBI patients age 16 or older who are at least one year post injury with stable cognitive deficits will be recruited

Exclusion Criteria:

* Had been treated with HBOT for any indiction prior to their inclusion.
* Have any other indication for HBOT
* Chest pathology incompatible with pressure changes
* Inner ear disease
* Patients suffering from claustrophobia.
* Inability to give written informed consent by the patient or his trustee.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-08; Primary Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Neurologic evaluation | 2 and 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Research & Development unit, Asaf-Harofeh Medical Center, Ẕerifin, Israel

REFERENCES:
- [Derived] Boussi-Gross R, Golan H, Fishlev G, Bechor Y, Volkov O, Bergan J, Friedman M, Hoofien D, Shlamkovitch N, Ben-Jacob E, Efrati S. Hyperbaric oxygen therapy can improve post concussion syndrome years after mild traumatic brain injury - randomized prospective trial. PLoS One. 2013 Nov 15;8(11):e79995. doi: 10.1371/journal.pone.0079995. eCollection 2013. PMID 24260334